CLINICAL TRIAL: NCT00294372
Title: Randomised, Double-blind, Placebo-controlled 7 Day Monotherapy Phase IIa Study to Evaluate the Antiviral Activity and Safety of Increasing Doses of Oral Administered RTV-boosted BILR 355 BS (75 mg and 150 mg Twice Daily) in HIV-1-infected, NNRTI-experienced Patients, Followed by 28 Day Combination Therapy With Tipranavir or Lopinavir Based HAART-regimen
Brief Title: Phase II Study on the Antiviral Activity and Safety of BILR 355 BS in HIV-1 Infected, NNRTI-treated Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1188.31
Record Dates: First submitted 2006-02-20; First posted 2006-02-22 (Estimated); Last update posted 2013-11-14 (Estimated); Status verified 2013-11

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Drug: BILR 355 BS
Drug: Placebo

SUMMARY:
The general aim is to evaluate the antiviral activity and safety of increasing doses of oral administered RTV-boosted BILR 355 BS (75 mg and 150 mg twice daily) in HIV-1-infected, NNRTI-experienced patients, followed by 28 day combination therapy with Tipranavir or Lopinavir based HAART-regimen

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent in accordance with GCP and local regulatory requirements prior to trial participation.
2. HIV-1 infected males or females >= 18 years of age.
3. History of NNRTI based HAART >= 8 weeks and at least one, but not more than 3 NNRTI-associated resistance mutations by current genotype
4. TPV/r or LPV/r susceptible
5. CD4+ T lymphocyte count >= 100 cells/?l.

7. HIV-1 viral load >= 2000 copies/mL at screening. 8. Karnofsky score >= 70 9. Based on the antiviral resistance profile of the patients virus, the investigator must be able to construct a background HAART treatment regimen (OBR) such that the patient will receive 3 effective ARV drugs, in addition to his study medication.

10. Acceptable screening laboratory values (Visit 1) that indicate adequate baseline organ function. Laboratory values are considered to be acceptable if the following apply: Absolute neutrophil count (ANC) >750/mm3 Hemoglobin >= 10 g/dL Platelet count >99,000/mm3 AST, ALT , and alkaline phosphatase < 2.5xULN >= DAIDS Grade 1) Total bilirubin <2.5xULN Serum amylase <1.5xULN 11. Acceptable medical history, as assessed by the investigator, with chest x-ray results and ECG within 1 year of study participation.

12. Willingness to abstain from ingesting substances which may alter plasma study drug levels by interaction with the cytochrome P450 system 13. A prior AIDS defining event, excluding mycobacterial and invasive fungal infections, is acceptable as long as it has resolved or the subject has been on stable treatment (e.g. opportunistic infection) for at least 12 weeks before screening (Visit 1). Note that prior oral thrush, candida esophagitis and cutaneous candida is acceptable.

Exclusion Criteria:

1. The following resistance mutations demonstrated at any time prior to starting trial therapy: V106A and/or Y188L
2. Female patients of child-bearing potential who:

   have a positive serum pregnancy test at screening or during the study, are breast feeding, are planning to become pregnant, are not willing to use a barrier method of contraception.
3. Active Hepatitis B or C disease defined as HBsAg positive or HCV RNA positive with AST/ALT > DAIDS Grade 1
4. Acute/previous mycobacterial or invasive fungal infection requiring therapy or prophylaxis with drugs interfering with or significantly affected by the cytochrome P450 system
5. Use of investigational medications within 30 days before study entry or during the trial.
6. Use of concomitant drugs that may significantly reduce plasma levels of the study medications.
7. Use of immunomodulatory drugs within 30 days before study entry or during the trial (e.g. interferon, cyclosporin, hydroxyurea, interleukin 2).
8. Patients currently treated with systemic ant-cancer chemotherapy
9. Inability to adhere to the requirements of the protocol, including active substance abuse, as defined by the investigator.
10. In the opinion of the investigator, likely survival of less than 12 months because of underlying disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36
Dates: Start 2006-02; Primary Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be reduction in plasma HIV-1 RNA from baseline to day 8, expressed in log10 copies/mm3. | day 8

SECONDARY OUTCOMES:
Virologic response at Day 8 and Day 35 using <400 copies/mL and 0.5, 1 and 1.5 log10 reduction in viral load from baseline | up to week 5
Change from baseline in viral load at each visit | up to week 9
Change from baseline in CD4+ cell counts at each visit | up to week 9
Time averaged change from baseline in viral load through Days 8 and 35 | up to week 5
Number of reverse transcriptase (RT) mutations at baseline | up to week 5
Number of NNRTI resistance-associated mutations at baseline (refer to Appendix 10.4) | up to week 5
The presence of specific RT mutations (both in the list of NNRTI mutations and not in the list for exploratory purposes) at baseline | up to week 5
The inhibitory quotient and minimum measured concentration of the analyte in plasma (Cmin) | up to Day 8
Exploration of mutations that emerge with exposure to BILR 355 BS to determine the effect on both viral load and IC50 fold change from reference | up to week 5
Area under the concentration-time curve of the analyte in plasma over the time interval 0 to 12 hours post-dose (AUC0-12h) | up to week 5
Maximum measured concentration of the analyte in plasma (Cmax) | up to week 5
Changes in total cholesterol, LDL, HDL and triglycerides from baseline to days 8 and 35 | up to week 9
Incidence of rash, hepatic events, and CNS adverse events | up to week 9
Incidence of any adverse events (treatment related and unrelated) | up to week 9
Incidence of laboratory test abnormalities | up to week 9
Incidence of serious adverse events (including AIDS-defining events) | up to week 9
Incidence of ≥ DAIDS 2 Grade elevation in ALT/AST | up to week 9
Incidence of AEs leading to discontinuation from the study | up to week 9

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — Boehringer Ingelheim
Locations (11):
- Germany (11):
  - Boehringer Ingelheim Investigational Site, Berlin
  - Boehringer Ingelheim Investigational Site, Bochum
  - Boehringer Ingelheim Investigational Site, Bonn
  - Boehringer Ingelheim Investigational Site, Erlangen
  - Boehringer Ingelheim Investigational Site, Frankfurt am Main
  - Boehringer Ingelheim Investigational Site, Hamburg
  - Boehringer Ingelheim Investigational Site, Hanover
  - Boehringer Ingelheim Investigational Site, Heidelberg
  - Boehringer Ingelheim Investigational Site, Mainz
  - Boehringer Ingelheim Investigational Site, München
  - Boehringer Ingelheim Investigational Site, Ulm